CLINICAL TRIAL: NCT03839303
Title: Infra-zygomatic Mini Implant Supported Appliance for Distalization and Intrusion of Maxillary Dentition Compared to Headgear in Growing Patients: A Randomized Clinical Trial
Brief Title: Comparison Between Mini Implant Supported Appliance and Headgear in Treatment of Maxillary Excess in Growing Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Khaled Mohamed Mohamed, Resident in orthodontic department of Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-11-1
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Class II Division 1 Malocclusion
MeSH Terms: conditions — Malocclusion, Angle Class II

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mini Implant Supported Appliance (Experimental): this group will receive an Infra-zygomatic Mini Implant Supported Appliance after leveling and alignment of the four upper incisors for 8 months or till class I canine or incisors realation is reached with follow up every month
  Interventions: Device: Infra-zygomatic Mini Implant Supported Appliance
- Headgear (Active Comparator): this group will receive a high pull headgear appliance attached to a removable acrylic maxillary splint for 8 months or till class I canine or incisors realation is reached with follow up every month
  Interventions: Device: high pull head gear

INTERVENTIONS:
Device: Infra-zygomatic Mini Implant Supported Appliance — 1. leveling and alignment of the four maxillary incisors
  2. infra zygomatic mini-implant will be placed bilaterally
  3. wire frame work that is designed resembling the inner bow of headgear will be adapted to the upper arch
  4. a heavy arch wire engaging the 4 incisors will be attached to the wire frame work
  5. orthopedic force will be delivered from the mini-implants to the wire frame work
  Arms: Mini Implant Supported Appliance
Device: high pull head gear — 1. acrylic maxillary splint is made with flying tubes
  2. high pull head gear is adapted to be inserted in the flying tubes
  Arms: Headgear

SUMMARY:
The aim of the study is to compare an Infra-zygomatic Mini implant supported appliance with headgear in distalization and intrusion of maxillary dentition for treatment of growing patients with class II malocclusion (maxillary excess)

DETAILED DESCRIPTION:
In this randomized trial, 2 groups will be included. The first group will receive an Infra-zygomatic Mini implant supported appliance. In the second group, the patient will receive a removable high pull headgear. the follow-up period will be 8 months or till class I canine or incisors relation is obtained. the assessment will be through a lateral cephalogram

ELIGIBILITY:
Inclusion Criteria:

1. Growing patients ( cervical vertebrae maturation stage cs2-cs3 )
2. Maxillary excess
3. Minimum overjet 4 mm
4. class II canines or incisors
5. Increased incisal show at rest and on smiling
6. Normal and increased vertical growth pattern
7. No previous orthodontic treatment
8. No congenitally messing teeth except third molars

Exclusion Criteria:

1. Inadequate incisal show
2. Class II with deficient mandible and normal maxilla
3. Patients with any syndrome
4. Patients with horizontal growth pattern

Ages: 7 Years to 15 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 26 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-11-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Anteroposterior position changes of upper first molars. | 8 months
  Measurements on the lateral cephalogram
Anteroposterior position changes of the maxilla | 8 months
  Measurements on the lateral cephalogram

SECONDARY OUTCOMES:
Vertical position changes in maxilla | 8 months
  Measurements on the lateral cephalogram
Vertical position changes of upper first molars | 8 months
  Measurements on the lateral cephalogram
Position changes of upper incisors | 8 months
  Measurements on the lateral cephalogram
Anteroposterior skeletal changes in mandible | 8 months
  Measurements on the lateral cephalogram

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Afifi, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided